CLINICAL TRIAL: NCT04681118
Title: Intermediate-size Patient Population Expanded Access Protocol: Repeated Administration of Nurown® (Autologous Mesenchymal Stem Cells Secreting Neurotrophic Factors) for the Treatment of Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Expanded Access Protocol: Repeated Administration of Nurown® (Autologous MSC-NTF Cells) for the Treatment of ALS
Status: No longer available | Type: Expanded Access
Sponsor: Brainstorm-Cell Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: BCT-003-US
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Biological: NurOwn (MSC-NTF cells) — Intrathecal administration

SUMMARY:
Expanded Access for treatment with investigational product MSC-NTF cells(NurOwn®) for participants who completed all scheduled treatments and follow-up assessments in the BCT-002-US study

DETAILED DESCRIPTION:
This is an Intermediate-size patient population Expanded Access Protocol (EAP) to provide NurOwn® (MSC-NTF cells) for eligible ALS participants who completed the BCT-002-US phase 3 ALS clinical trial and have received all three IT treatments.

The participants will undergo up to three intrathecal (IT) treatments with NurOwn® (MSC-NTF cells).

In the first treatment period, the participant received up to three intrathecal (IT) treatments with NurOwn® (MSC-NTF cells) at T1, T2 and T3 and was followed for 12 weeks after the third treatment.

In the second treatment period, the participant will receive up to three intrathecal (IT) treatments with NurOwn® (MSC-NTF cells) every 8 weeks at T4, T5 and T6.

Following the last EAP treatment, the participant will be followed for three additional monthly visits (in-person, if feasible, or by telephone call or telemedicine in consideration of the ongoing COVID-19 pandemic) through the final protocol visit, during which the ALSFRS-R and safety assessments will be collected

ELIGIBILITY:
Inclusion Criteria:

1. Participation in the BCT-002-US study, successful completion of all scheduled treatments and follow-up assessments.

2 Able to provide to the Investigator written informed consent regarding the investigational drug, or, as applicable, on whose behalf a legally authorized representative of the participant has provided such consent.

3. Able to safely undergo all study procedures.

Exclusion Criteria:

1. Inability to lie flat for the duration of intrathecal cell transplantation and/or bone marrow biopsy, or inability to tolerate treatment procedures for any other reason (lying flat with BiPAP or NIV are not exclusionary).
2. History of clinically significant autoimmune disease (excluding thyroid disease) myelodysplastic or myeloproliferative disorder, leukemia or lymphoma, whole body irradiation, hip fracture, or severe scoliosis.
3. Any unstable clinically significant medical condition other than ALS (e.g., within six months of baseline, had myocardial infarction, angina pectoris, and/or congestive heart failure), treatment with anticoagulants that, in the opinion of the Investigator, would compromise the safety of the participant.
4. Any history of malignancy within the previous 5 years, with the exception of non- melanoma localized skin cancers (with no evidence of metastasis, significant invasion, or re-occurrence within three years of baseline).
5. Current use of immunosuppressant medication or use of such medication within 4 weeks of the pre-treatment visit.
6. Any history of acquired or inherited immune deficiency syndrome.
7. Tracheostomy and/or mechanical ventilation. Feeding tube use, BiPAP or NIV are not exclusionary.
8. Pregnant women or women currently breastfeeding or unwilling to use effective birth control methods during the treatment (if of childbearing age).
9. Positive test result for Hepatitis B virus (HBV; surface antigen (HBsAg) and IgM antibodies to core antigen (IgM anti-HBc)), Hepatitis C virus (HCV), Human Immune deficiency virus (HIV) 1 and 2.

Ages: 18 Years to 63 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California Irvine Alpha Stem Cell Clinic, Irvine, California
  - California Pacific Medical Center, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Medical School, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota